CLINICAL TRIAL: NCT05656534
Title: Orexin Receptor Antagonists as Modulators of Threat Sensitivity in Individuals With Alcohol Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Stephanie M Gorka, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022H0265; 1R21AA030097-01A1 (NIH)
Record Dates: First submitted 2022-12-11; First posted 2022-12-19 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder
Keywords: suvorexant; alcohol use disorder; electromyography; functional magnetic resonance imaging
MeSH Terms: conditions — Alcoholism | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Individuals will take a placebo pill during the Acute Drug Challenge and daily for 28 days.
  Interventions: Other: Placebo
- Suvorexant Treatment (Experimental): Individuals will take 10mg of suvorexant (Merck & Co Inc.) during the Acute Drug Challenge and daily for 28 days.
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG, fMRI). Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. After the pre-treatment visits participants will take one pill of SUV at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete an EMG. Laboratory assessments will occur during peak concentration, 2 hours post-ingestion. At the end of the visit, participants will be given a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side effects and potential drug-drug interactions. At the end of the 28 days, participants will complete post-treatment lab visits.
  Other Names: Belsomra
  Arms: Suvorexant Treatment
Other: Placebo — This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG, fMRI). The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visits, participants will take one pill at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete the EMG paradigm. At the end of the visit participants will be provided a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side. At the end of the 28 days, participants will complete post-treatment lab visits.
  Arms: Control

SUMMARY:
The goal of this double-blind clinical trial is to further explore if, how, and for whom orexin antagonism modifies brain-behavior stress targets in moderate to severe alcohol use disorder (AUD). The main questions it aims to answer are:

* Does an acute dose of suvorexant (SUV) and/or daily use of SUV modify brain-behavior targets of AUD dysfunction?
* Does daily SUV use change alcohol behavior and if so, is this change in behavior linked to brain-behavior change?

Participants will be randomized to a treatment group (SUV or placebo) and protocol arm, electromyography (EMG) only or EMG+functional magnetic resonance imaging (fMRI). Participants will be asked to complete the following:

* Baseline lab visit(s) that include the psychophysiological stress paradigm (EMG only or EMG+fMRI, dependent upon randomization).
* Acute drug challenge where the participant will return to the lab to repeat the stress paradigm following administration of a single dose of either 10mg SUV or placebo.
* Medication trial where participants will be instructed to take 10mg capsules of SUV or placebo orally each night before bedtime for 4-weeks.
* Daily reports of medication adherence, side-effects, sleep, alcohol use, and mood will be collected via smartphones during the 4-week medication trial.
* Post-treatment lab visit(s) where participants will return to the lab at the end of the medication trial and complete the same stress paradigm from baseline (EMG only or EMG+fMRI, dependent upon randomization).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Participant is able to give informed consent.
* Generally medically and physically healthy as confirmed by medical history.
* Meet DSM-5 diagnostic criteria for current moderate or severe AUD.
* Engage in heavy alcohol use defined as drinking equal or greater than 14 standard drinks per week if male and equal or greater than 7 standard drinks per week if female.

Exclusion Criteria:

* Clinically significant medical or neurological condition (e.g., liver disease, narcolepsy, complex sleep behaviors, severe hepatic impairment, COPD, severe obstructive sleep apnea).
* Current cognitive dysfunction (traumatic brain injury, mental retardation, organic mental syndrome, pervasive developmental disorder, or dementia).
* Current use of antihistamines, strong or moderate inhibitors of CYP3A liver enzymes, strong CYP3A inducers, or digoxin.
* Current or past DSM-5 diagnosis of mania, schizophrenia, psychosis, suicidality, major depressive disorder, or obsessive compulsive disorder.
* Current substance use disorder other than alcohol or mild cannabis use disorder.
* Treatment seeking for AUD.
* Recent psychotropic medication use in the past 2 months.
* Currently smokes 5 or more cigarettes (or electronic equivalent) per day.
* BMI equal or greater than 35.
* Engage in night-shift work.
* Lack of fluency in English.
* Presence of ferrous-containing metal in the body.
* Inability to tolerate small, enclosed spaces.
* Deafness in one or both ears.
* Currently pregnant (positive pregnancy test), lactating, or not agreeing to use birth control methods during the duration of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including fMRI, startle eyeblink, and behavior, from this project will be submitted to the NIAAA Data Archive (NDA) at the subject level along with appropriate supporting documentation to enable efficient use of the data by the research community. We will follow instructions as discussed in the NIAAA Data Archive Data Sharing Terms and Conditions.
  We will follow the two-tier procedure described in the guidelines:
  1. Raw continuous fMRI recordings will be submitted in standard formats (Matlab mat format, DICOM format and NIFTI format). Experimental condition information will be supplied in text format along with other critical information.
  2. Analyzed data (BOLD data, BOLD-startle eyeblink data) associated with a manuscript will be shared as soon as possible, and at the latest, at the time of publication of the manuscript. These data may be accompanied, if applicable, by other data such as behavioral data, supplied in text format.
Time Frame: The data, as outlined above, will be submitted to the NIAAA Data Archive biannually per NIAAA requirements throughout the duration of the study.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via print advertisements, word-of-mouth referrals, and internet postings throughout Columbus and the surrounding area between November 2022 and June 2024. The first participant was enrolled on November 29th, 2022 and the last participant was enrolled in June 2024.
Pre-assignment Details: Of 81 enrolled participants, 64 participants were randomized to treatment.
Groups:
- Placebo+EMG Only: Individuals will take a placebo pill during the Acute Drug Challenge and daily for 28 days.
  Placebo: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG only). The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visits, participants will take one pill at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete the EMG paradigm. At the end of the visit participants will be provided a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side. At the end of the 28 days, participants will complete post-treatment lab visits.
- Suvorexant+EMG Only: Individuals will take 10mg of suvorexant (Merck & Co Inc.) during the Acute Drug Challenge and daily for 28 days.
  Suvorexant: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG only). Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. After the pre-treatment visits participants will take one pill of SUV at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete an EMG. Laboratory assessments will occur during peak concentration, 2 hours post-ingestion. At the end of the visit, participants will be given a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side effects and potential drug-drug interactions. At the end of the 28 days, participants will complete post-treatment lab visits.
- Placebo+fMRI+EMG: Individuals will take a placebo pill during the Acute Drug Challenge and daily for 28 days.
  Placebo: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG +fMRI). The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visits, participants will take one pill at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete the EMG paradigm. At the end of the visit participants will be provided a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side. At the end of the 28 days, participants will complete post-treatment lab visits.
- Suvorexant+fMRI+EMG: Individuals will take 10mg of suvorexant (Merck & Co Inc.) during the Acute Drug Challenge and daily for 28 days.
  Suvorexant: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG, fMRI). Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. After the pre-treatment visits participants will take one pill of SUV at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete an EMG. Laboratory assessments will occur during peak concentration, 2 hours post-ingestion. At the end of the visit, participants will be given a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side effects and potential drug-drug interactions. At the end of the 28 days, participants will complete post-treatment lab visits.
Period: Overall Study
Arm/Group | Placebo+EMG Only | Suvorexant+EMG Only | Placebo+fMRI+EMG | Suvorexant+fMRI+EMG
Started | 18 | 18 | 15 | 13
Completed | 16 | 16 | 15 | 13
Not Completed | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo + EMG Only: Individuals will take a placebo pill during the Acute Drug Challenge and daily for 28 days.
  Placebo: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG only). The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visits, participants will take one pill at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete the EMG paradigm. At the end of the visit participants will be provided a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side. At the end of the 28 days, participants will complete post-treatment lab visits.
- Suvorexant + EMG Only: Individuals will take 10mg of suvorexant (Merck & Co Inc.) during the Acute Drug Challenge and daily for 28 days.
  Suvorexant: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG only). Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. After the pre-treatment visits participants will take one pill of SUV at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete an EMG. Laboratory assessments will occur during peak concentration, 2 hours post-ingestion. At the end of the visit, participants will be given a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side effects and potential drug-drug interactions. At the end of the 28 days, participants will complete post-treatment lab visits.
- Placebo+fMRI+EMG: Individuals will take a placebo pill during the Acute Drug Challenge and daily for 28 days.
  Placebo: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG, fMRI). The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visits, participants will take one pill at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete the EMG paradigm. At the end of the visit participants will be provided a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side. At the end of the 28 days, participants will complete post-treatment lab visits.
- Total: Total of all reporting groups
Arm/Group | Placebo + EMG Only | Suvorexant + EMG Only | Placebo+fMRI+EMG | Suvorexant+fMRI+EMG | Total
Number analyzed (Participants) | 18 | 18 | 15 | 13 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 15 | 13 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 8 | 37
  Male | 8 | 8 | 6 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 2 | 6
  Not Hispanic or Latino | 17 | 15 | 15 | 11 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 3
  White | 18 | 13 | 15 | 12 | 58
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Startle Eyeblink Electromyographic (EMG) Response to Stress With an Acute Dose of Suvorexant
Description: Startle EMG responses were collected during the well-validated No-Predictable-Unpredictable threat paradigm. The task includes within-subjects conditions and raw EMG responses were averaged for each condition. To quantify the difference between threat and no-threat periods, we calculated a standardized residual score for unpredictable threat (U-threat) by saving the variance leftover (i.e., the amount of variability in a dependent variable [DV] that is not explained by an independent variable [IV]) in a simple linear regression, where the no-threat EMG startle average (IV) was entered to predict the U-threat EMG startle average (DV). The U-threat residual score was used as the primary variable. It has a mean of zero and higher scores reflect greater startle reactivity to U-threat. U-threat residual scores were calculated for the baseline session and the acute challenge.
Time Frame: Change from baseline to 2 hours post-ingestion of an acute dose of suvorexant.
Population: A total of 57 participants were included. Missing data was due to attrition, poor quality startle eyeblink data, or technical errors during startle data collection.
Measure: Mean (Standard Error); unit: Standardized residual scores
Arm/Group | Control | Suvorexant Treatment
Number analyzed (Participants) | 30 | 27
Standardized residual scores
  Pre-Treatment Startle to U-threat | 0.01 (0.18) | .24 (0.19)
  Acute Challenge Startle to U-threat | 0.01 (0.17) | -0.18 (0.18)
Statistical Analysis 1: Comparison: Control vs Suvorexant Treatment; Test type: Superiority; p = .19, ANOVA; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.20 to 1.10], Standard Error of Mean 0.31

2. Primary Outcome: Startle Eyeblink Electromyographic (EMG) Response to Stress With Daily Use of Suvorexant.
Description: Startle EMG responses were collected during the well-validated No-Predictable-Unpredictable threat paradigm. The task includes within-subjects conditions and raw EMG responses were averaged for each condition. To quantify the difference between threat and no-threat periods, we calculated a standardized residual score for unpredictable threat (U-threat) by saving the variance leftover (i.e., the amount of variability in a dependent variable [DV] that is not explained by an independent variable [IV]) in a simple linear regression, where the no-threat EMG startle average (IV) was entered to predict the U-threat EMG startle average (DV). The U-threat residual score was used as the primary variable. It has a mean of zero and higher scores reflect greater startle reactivity to U-threat.
Time Frame: Change from baseline to post-treatment, up to 2 months.
Population: A total of 54 participants were included. Missing data was due to attrition, poor quality startle eyeblink data, or technical errors during startle data collection.
Measure: Mean (Standard Error); unit: Standardized residual scores
Arm/Group | Control | Suvorexant Treatment
Number analyzed (Participants) | 29 | 25
Standardized residual scores
  Pre-Treatment Startle to U-threat | -0.13 (0.14) | 0.28 (0.18)
  Post-treatment Startle to U-threat | 0.08 (0.19) | -0.23 (0.14)
Statistical Analysis 1: Comparison: Control vs Suvorexant Treatment; We conducted a repeated measures analysis of variable with session (pre-treatment vs. post-treatment) as a within-subjects variable and treatment arm as a between-subjects variable. Standardized residual scores reflecting startle reactivity to unpredictable threat (> no-threat) was the dependent variable; Test type: Superiority; p = 0.03, ANOVA; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.07 to 1.38], Standard Error of Mean 0.33

3. Primary Outcome: Percentage of Heavy Drinking Days During Daily Use of Suvorexant.
Description: Percentage of heavy drinking days (PHDD) was calculated each week for all four weeks of the trial. A heavy drinking day was defined using NIH criteria: 5+ drinks for males and 4+ drinks for females in a single day. We conducted a multilevel mixed model with PHDD from week 1 to 4 as the within-subjects variable and treatment arm as the between subjects variable.
Time Frame: Change from baseline to post-treatment, over the course of 4 weeks.
Population: All 64 participants randomized to treatment were analyzed.
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Control | Suvorexant Treatment
Number analyzed (Participants) | 33 | 31
percentage of heavy drinking days
  Week 1 PHDD | 27.7 (4.0) | 29.5 (3.6)
  Week 2 PHDD | 31.2 (3.6) | 29.5 (3.9)
  Week 3 PHDD | 27.2 (4.2) | 24.4 (3.1)
  Week 4 PHDD | 27.6 (3.3) | 16.9 (2.6)
Statistical Analysis 1: Comparison: Control vs Suvorexant Treatment; Test type: Superiority; p = .01, Mixed Models Analysis

4. Secondary Outcome: Changes in Neural Activation During Unpredictable Stress Anticipation Following Daily Use of Suvorexant.
Description: Activation parameter estimates (arbitrary units) were extracted from anatomical bilateral aINS masks for each individual, pre and post treatment. Specifically, activation parameter estimates were extracted from anticipation of unpredictable threat > anticipation of no-threat individual contrast maps for each scanning session. Greater values reflect greater activation in the bilateral insula during the anticipation of unpredictable threat. A repeated measures analysis of variance was used to test the session (time 1 vs. time 2) by treatment arm interaction on bilateral aINS activation during unpredictable threat. Significance was set at p <.05
Time Frame: Change from baseline to post-treatment, up to 2 months.
Population: A subset of participants were randomized to complete functional magnetic resonance imaging (fMRI) pre- and post-treatment. Only individuals with two scanning sessions were analyzed.
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | Control | Suvorexant Treatment
Number analyzed (Participants) | 13 | 13
arbitrary units
  Pre-Treatment Bilateral aINS | 0.330 (0.141) | 0.652 (0.141)
  Post-Treatment Bilateral aINS | 0.482 (0.153) | 0.226 (0.153)
Statistical Analysis 1: Comparison: Control vs Suvorexant Treatment; A session (pre vs. post) by treatment arm (suvorexant vs. placebo) repeated measures analysis of variance (ANOVA) was performed. The effect of session was then probed within each treatment arm; Test type: Superiority; p < .05, ANOVA; Repeated measures ANOVA modeling session (pre. vs. post) by treatment arm; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.01 to 1.20], Standard Error of Mean 0.28

ADVERSE EVENTS:
Time Frame: 2 months.
Groups:
- Suvorexant+fMR+EMG: Individuals will take 10mg of suvorexant (Merck & Co Inc.) during the Acute Drug Challenge and daily for 28 days.
  Suvorexant: This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment lab visits (EMG, fMRI). Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. After the pre-treatment visits participants will take one pill of SUV at the Acute Drug Challenge under medical supervision. Ninety minutes post ingestion participants will complete an EMG. Laboratory assessments will occur during peak concentration, 2 hours post-ingestion. At the end of the visit, participants will be given a blister pack with 28 pills. Participants will be instructed to take one pill orally about 30 minutes prior to sleep time each night for 28 days. Participants will be provided education about common side effects. Participants will complete daily surveys to monitor side effects and potential drug-drug interactions. At the end of the 28 days, participants will complete post-treatment lab visits.
Arm/Group | Placebo + EMG Only | Suvorexant + EMG Only | Placebo+fMRI+EMG | Suvorexant+fMR+EMG
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 3/18 | 3/18 | 3/15 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + EMG Only (N=18) | Suvorexant + EMG Only (N=18) | Placebo+fMRI+EMG (N=15) | Suvorexant+fMR+EMG (N=13)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Disturbances (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT05656534/Prot_SAP_000.pdf